CLINICAL TRIAL: NCT05430880
Title: Study of the Performance of VCO2 Variation as an Indicator of Fluid Responsiveness in Intensive Care Unit
Brief Title: Cardiac Responsiveness Assessment by CO2
Acronym: CRAC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 485
Record Dates: First submitted 2022-06-20; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: VCO2 Variation in Intensive Care as a Marker of Fluid Responsiveness; Cardiac Index Variation Transpulmonary Thermodilution in Patients on Controlled Ventilation With Shock
Keywords: cardiac output; VCO2; fluid responsiveness; Intensive care unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "CRAC" patients : ICU patients ventilated and shocked: Patient hospitalized in intensive care.
  Patient sedated and mechanically ventilated in Volume Assisted Controlled mode.
  Patient with hypotension (MAP <65 mmHg OR SAP <90 mmHg) AND / OR under continuous infusion of Norepinephrine / Dobutamine / Epinephrine
  Patient equipped with a cardiac output measurement system by transpulmonary thermodilution (PICCO®) with a femoral arterial module; as well as a central venous route in the superior vena cava territory.
  Inclusion after agreement of the patient or his trusted person after validation of the inclusion criteria and verification of the absence of exclusion criteria.
  Interventions: Diagnostic Test: impact of fluid challenge on the cardiac index and CO2 respiratory parameters analysis (VCO2, EtCO2)

INTERVENTIONS:
Diagnostic Test: impact of fluid challenge on the cardiac index and CO2 respiratory parameters analysis (VCO2, EtCO2) — Preliminary daily data will record: demographic, ventilatory (tidal volume, FiO2, positive expiratory pressure, compliance, respiratory rate, I/E ratio) and biological parameters (fibrinogen, CRP, leukocytes count, PaO2, PvO2, PaCO2, PvCO2, CO2gap, arterial lactate, ScvO2, platelets count)
  1. st step CO2 record (between Time-6minutes and T0; T0 corresponding to fluid challenge) VCO2 and EtCO2 (End-tidal CO2) automated measurement by Hamilton module. Average VCO2 obtained before fluid challenge.
     CI (cardiac index): measurement by calibration of the PiCCO module with 3 cold boli.
  2. nd step: Crystalloid (ringer lactate) filling 500mL in 5 minutes
  3. rd step CO2 record (between T+5min and Time+11minutes): VCO2 and EtCO2: automated measurement by Hamilton module. Average VCO2 obtained after fluid challenge.
  CI (cardiac index): measurement by calibration of the PiCCO module with 3 cold boli

SUMMARY:
The increase of cardiac output resulting from increased blood volume (systolic ejection volume) during intravenous fluid administration defines a state of fluid responsiveness.

Fluid responsiveness in intensive care patients with circulatory failure (shock) needs to be carefully evaluated because only half of the patients are fluid responsive and excessive fluid administration is harmful.

To reliably assess this state, it is currently necessary to perform either invasive cardiac output monitoring or ultrasound evaluation before and after a fluid administration (called fluid challenge). It is either an invasive procedure or a time-consuming technique (that might depend on operator experience and patient echogenicity).

The investigators foresee a potential benefit for an objective quick-answering screening tool that does not require additional monitoring.

Instantaneous CO2 production rate (VCO2) calculated automatically by the most recent ventilators (Hamilton C5-C6) via the analysis of exhaled gases.

There is an established physiological link between cardiac output, arterial oxygen transport to cells and CO2 production by cell metabolism.

The variation in End-Tidal CO2 (another parameter derived from exhaled CO2) is conventionally monitored in the operating room; it can show sudden changes in cardiac output. In intensive care, the EtCO2 variation is probably less sensitive than the variation in VCO2 to detect changes in cardiac output.

The aim of this study is to show that the variation in VCO2 as shown on ventilators during a fluid challenge test has satisfactory diagnostic performance in the detection of fluid responsiveness in patients with circulatory failure in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in intensive care.
* Patient sedated and mechanically ventilated in Volume Assisted Controlled mode.
* Patient with hypotension (MAP <65 mmHg OR SAP <90 mmHg) AND / OR under continuous infusion of Norepinephrine / Dobutamine / Epinephrine
* Patient equipped with a cardiac output measurement system by transpulmonary thermodilution (PICCO®) with a femoral arterial module; as well as a central venous route in the superior or inferior vena cava territory.

Exclusion Criteria :

* Patient under 18 years old
* Patient under guardianship without the possible consent of the guardian
* Pregnant woman
* Pathologies and maneuvers strongly affecting CO2 purification: Diagnosed pulmonary embolism, Prone positioning for less than 60 minutes, Exogenous intake of sodium bicarbonate less than 60 minutes ago (with the exception of an renal replacement therapy in place for more than 60 minutes)
* Recent change in respiratory quotient: Change in enteral or parenteral nutrition solution for less than 3 hours
* Pathology affecting CO2 metabolism: Fever> 39 ° c, Intense chills.
* Patients with unstable ventilation over the hour before inclusion.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study concerns adult subjects in intensive care with a state of circulatory failure (shock), in whom the indication of fluid vascular filling is to be discussed.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
The main endpoint is the performance of the variation of the VCO2 (noted ΔVCO2 after obtaining an average before vascular filling VCO2m1 and an average after vascular filling VCO2m2) in ml/min in the detection of fluid-responsiveness. | at the inclusion during less than fifteen minutes
  The investigators will analyze the VCO2 variation performance to detect fluid responsiveness as established by the sensitivity, specificity, positive and negative predictive values as well as by analysis of the ROC curve. The Gold Standard used as a comparator for this test is the change in cardiac index (ΔIC in L/min/m2) measured by transpulmonary thermodilution before / after fluid challenge and considered significant if greater than or equal to 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Anesthésie-réanimation, Lyon, France